CLINICAL TRIAL: NCT04330989
Title: UNCPMZ 41901 - An Integrated Strategy to Support Antiretroviral Therapy and Pre-exposure Prophylaxis Adherence for HIV Prevention in Pregnant and Breastfeeding Women: a Pilot Study
Brief Title: An Integrated Strategy to Support Antiretroviral Therapy and Pre-exposure Prophylaxis Adherence for HIV Prevention in Pregnant and Breastfeeding Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-1060; R01AI131060 (NIH); UNCPMZ 41901 (Other: UNC)
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Results first posted 2023-01-09 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-01

CONDITIONS: HIV-1-infection; Antenatal Care
Keywords: HIV Transmission; Antiretroviral Treatment; Pre-exposure Prophylaxis; Patient-centered Counseling; Adherence Supporter Training; Antenatal Care; HIV

STUDY DESIGN:
Intervention Model Description: This is a parallel pilot randomized trial in which participants randomly assigned to the control arm will receive antiretroviral adherence support about HIV treatment and prevention. Those randomized to the intervention arm will additionally receive a multi-component support strategy comprising integrated next-step counseling (iNSC) and adherence supporter training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group 1a: iNSC and Adherence supporter training (Experimental): HIV-positive women randomly assigned to the intervention arm will receive a multi-component support strategy comprising iNSC and adherence supporter training for ART.
  Interventions: Behavioral: iNSC and Adherence supporter training
- Group 1b: Standard of Care (No Intervention): HIV-positive participants randomly assigned to the control arm will antiretroviral educational material about HIV prevention and treatment (as appropriate to this arm).
- Group 2a: iNSC and Adherence supporter training (Experimental): HIV-negative women randomly assigned to the intervention arm will receive a multi-component support strategy comprising iNSC and adherence supporter training for PrEP.
  Interventions: Behavioral: iNSC and Adherence supporter training
- Group 2b: Standard of Care (No Intervention): HIV-negative participants randomly assigned to the control arm will receive educational material about HIV prevention and treatment (as appropriate to this arm).

INTERVENTIONS:
Behavioral: iNSC and Adherence supporter training — Integrated next step counseling: iNSC is a structured, patient-centered approach informed by motivational interviewing techniques, which aims to foster an environment for joint-problem solving in order that the participant may identify their individual needs to increase or sustain sexual health through biomedical and non-biomedical approaches. iNSC frames the counselling sessions as a non-judgmental discussion to explore the facilitators and challenges to sexual health and medication adherence.
  Adherence supporter training: Participants will be asked to identify a partner, family member, or friend to whom they are willing to disclose their HIV status (for HIV-positive women) or their intent to initiate PrEP (for HIV-negative women). Participants may also select a clinic-based peer to serve this adherence supporter role. Trainings will emphasize basic HIV knowledge, importance of antiretroviral adherence, potential drug side effects, and practical strategies for supporting adherence.
  Arms: Group 1a: iNSC and Adherence supporter training; Group 2a: iNSC and Adherence supporter training

SUMMARY:
This study is composed of two parallel, pilot randomized groups that will obtain preliminary data about the the acceptability, fidelity, and clinical outcomes associated with a multi-component adherence support strategy for HIV treatment and prevention among pregnant and breastfeeding women. The study will take place in Lilongwe, Malawi.

DETAILED DESCRIPTION:
If the anticipated gains for the prevention of mother-to-child HIV transmission (PMTCT) programs are to be realized, adherence to antiretroviral regimens will be critical. To date, however, there are few evidence-based approaches that are scalable and sustainable in busy, programmatic settings where HIV burden is high. The study seeks to implement the intervention, which includes patient-centered counseling and adherence supporter training, for both HIV-positive (for antiretroviral therapy, or ART) and HIV-negative (for pre-exposure prophylaxis, or PrEP) pregnant and breastfeeding women, thus providing a universal approach to support PMTCT programs holistically. The study will enroll pregnant women 18 years of age or older receiving antenatal care services at one of the designated study facilities. In Group 1, the study will enroll 100 HIV-positive women who started (or re-started, after a 6 months or longer treatment interruption) a first-line ART regimen within the past 30 days. In Group 2, the study will enroll 200 HIV-negative women willing to initiate and continue oral PrEP, in the form of tenofovir disoproxil fumarate and emtricitabine (TDF-FTC), and who report factors that place them at elevated risk for HIV acquisition.

ELIGIBILITY:
Eligibility criteria for enrollment in Group 1 (HIV-positive women):

Inclusion Criteria:

* Documented pregnancy by urine pregnancy test or physical exam
* Documented positive HIV status
* Initiated on first-line antiretroviral therapy (ART) within the past 30 days, either for the first time or after treatment interruption of 6 months or longer (if previously started but stopped ART)
* Willingness to remain in the study site's catchment area over the course of study follow-up and to comply with visit schedule
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Risk for intimate partner violence or social harms as a result of participation, in the judgement of the study personnel
* Other conditions that, in the judgment of the study personnel, would make participation in the study inappropriate

Eligibility criteria for enrollment in Group 2 (HIV-negative women):

Inclusion Criteria:

* Documented pregnancy by urine pregnancy test or physical exam
* Documented negative HIV status within the past three months
* Identified factor(s) for elevated risk for HIV acquisition, such as known positive or unknown partner HIV status; report of secondary sexual partners over the past 12 months; diagnosis of sexually transmitted infection over the past 12 months; use of post-exposure prophylaxis in the past 12 months; reported use of shared injection material or equipment; and/or unspecified concern about HIV acquisition during pregnancy and breastfeeding
* Willingness to initiate and continue HIV pre-exposure prophylaxis (PrEP) over the course of study follow-up
* Willingness to remain in the study site's catchment area over the course of study follow-up and to comply with visit schedule
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Positive HIV test at time of screening
* Positive hepatitis B surface antigen test at time of screening
* Renal insufficiency, defined as creatinine clearance <90 mL/min, history of known renal parenchymal disease, or known single kidney at time of screening
* Risk for intimate partner violence or social harms as a result of participation, in the judgement of the study personnel
* Other conditions that, in the judgment of the study personnel, would make participation in the study inappropriate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Chi, MD, MSc, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Bwaila District Hospital, Lilongwe, Malawi

REFERENCES:
- [Derived] Mutale W, Graybill LA, Saidi F, Phanga T, Amico KR, Freeborn K, Rosenberg NE, Hill LM, Hamoonga T, Richardson BD, Mollan KR, Chi BH. Evaluation of a combination adherence strategy to support HIV antiretroviral therapy for pregnancy and breastfeeding in Malawi: A pilot randomized clinical trial. PLoS One. 2025 Apr 28;20(4):e0319735. doi: 10.1371/journal.pone.0319735. eCollection 2025. PMID 40293995
- [Derived] Chi BH, Saidi F, Graybill LA, Phanga T, Mollan KR, Amico KR, Freeborn K, Rosenberg NE, Hill LM, Hamoonga T, Richardson B, Kalua T, Phiri S, Mutale W. A Patient-Centered, Combination Intervention to Support Adherence to HIV Pre-exposure Prophylaxis During Pregnancy and Breastfeeding: A Randomized Pilot Study in Malawi. J Acquir Immune Defic Syndr. 2024 Jan 1;95(1):42-51. doi: 10.1097/QAI.0000000000003309. PMID 37757844
- [Derived] Saidi F, Mutale W, Freeborn K, Rosenberg NE, Graybill LA, Maman S, Amico KR, Mollan KR, Phanga T, Milala B, Hill LM, Gottwalt AM, Phiri S, Kalua T, Chi BH. Combination adherence strategy to support HIV antiretroviral therapy and pre-exposure prophylaxis adherence during pregnancy and breastfeeding: protocol for a pair of pilot randomised trials. BMJ Open. 2021 Jun 30;11(6):e046032. doi: 10.1136/bmjopen-2020-046032. PMID 34193491

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1a: Integrated Next Step Counseling (iNSC) and Adherence Supporter Training: HIV-positive women randomly assigned to the intervention arm will receive a multi-component support strategy comprising Integrated Next Step Counseling (iNSC) and adherence supporter training for antiretroviral therapy (ART).
  iNSC and Adherence supporter training: Integrated next step counseling: iNSC is a structured, patient-centered approach informed by motivational interviewing techniques, which aims to foster an environment for joint-problem solving in order that the participant may identify their individual needs to increase or sustain sexual health through biomedical and non-biomedical approaches. iNSC frames the counselling sessions as a non-judgmental discussion to explore the facilitators and challenges to sexual health and medication adherence.
  Adherence supporter training: Participants will be asked to identify a partner, family member, or friend to whom they are willing to disclose their HIV status (for HIV-positive women) or their intent to initiate PrEP (for HIV-negative women). Participants may also select a clinic-based peer to serve this adherence supporter role. Trainings will emphasize basic HIV knowledge, importance of antiretroviral adherence, potential drug side effects, and practical strategies for supporting adherence.
- Group 2a: iNSC and Adherence Supporter Training: HIV-negative women randomly assigned to the intervention arm will receive a multi-component support strategy comprising Integrated Next Step Counseling (iNSC) and adherence supporter training for HIV pre-exposure prophylaxis (PrEP).
  iNSC and Adherence supporter training: Integrated next step counseling: iNSC is a structured, patient-centered approach informed by motivational interviewing techniques, which aims to foster an environment for joint-problem solving in order that the participant may identify their individual needs to increase or sustain sexual health through biomedical and non-biomedical approaches. iNSC frames the counselling sessions as a non-judgmental discussion to explore the facilitators and challenges to sexual health and medication adherence.
  Adherence supporter training: Participants will be asked to identify a partner, family member, or friend to whom they are willing to disclose their HIV status (for HIV-positive women) or their intent to initiate PrEP (for HIV-negative women). Participants may also select a clinic-based peer to serve this adherence supporter role. Trainings will emphasize basic HIV knowledge, importance of antiretroviral adherence, potential drug side effects, and practical strategies for supporting adherence.
Period: Overall Study
Arm/Group | Group 1a: Integrated Next Step Counseling (iNSC) and Adherence Supporter Training | Group 1b: Standard of Care | Group 2a: iNSC and Adherence Supporter Training | Group 2b: Standard of Care
Started | 51 | 49 | 100 | 100
Liveborn Infants During Study | 43 | 46 | 87 | 90
Completed | 41 | 43 | 88 | 83
Not Completed | 10 | 6 | 12 | 17

BASELINE CHARACTERISTICS:
Groups:
- Group 1a: iNSC and Adherence Supporter Training: HIV-positive women randomly assigned to the intervention arm will receive a multi-component support strategy comprising iNSC and adherence supporter training for ART.
  iNSC and Adherence supporter training: Integrated next step counseling: iNSC is a structured, patient-centered approach informed by motivational interviewing techniques, which aims to foster an environment for joint-problem solving in order that the participant may identify their individual needs to increase or sustain sexual health through biomedical and non-biomedical approaches. iNSC frames the counselling sessions as a non-judgmental discussion to explore the facilitators and challenges to sexual health and medication adherence.
  Adherence supporter training: Participants will be asked to identify a partner, family member, or friend to whom they are willing to disclose their HIV status (for HIV-positive women) or their intent to initiate PrEP (for HIV-negative women). Participants may also select a clinic-based peer to serve this adherence supporter role. Trainings will emphasize basic HIV knowledge, importance of antiretroviral adherence, potential drug side effects, and practical strategies for supporting adherence.
- Group 2a: iNSC and Adherence Supporter Training: HIV-negative women randomly assigned to the intervention arm will receive a multi-component support strategy comprising iNSC and adherence supporter training for PrEP.
  iNSC and Adherence supporter training: Integrated next step counseling: iNSC is a structured, patient-centered approach informed by motivational interviewing techniques, which aims to foster an environment for joint-problem solving in order that the participant may identify their individual needs to increase or sustain sexual health through biomedical and non-biomedical approaches. iNSC frames the counselling sessions as a non-judgmental discussion to explore the facilitators and challenges to sexual health and medication adherence.
  Adherence supporter training: Participants will be asked to identify a partner, family member, or friend to whom they are willing to disclose their HIV status (for HIV-positive women) or their intent to initiate PrEP (for HIV-negative women). Participants may also select a clinic-based peer to serve this adherence supporter role. Trainings will emphasize basic HIV knowledge, importance of antiretroviral adherence, potential drug side effects, and practical strategies for supporting adherence.
- Total: Total of all reporting groups
Arm/Group | Group 1a: iNSC and Adherence Supporter Training | Group 1b: Standard of Care | Group 2a: iNSC and Adherence Supporter Training | Group 2b: Standard of Care | Total
Number analyzed (Participants) | 51 | 49 | 100 | 100 | 300
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [23 to 30] | 27 [24 to 33] | 25 [22 to 28] | 24 [21 to 28] | 25 [22 to 29]
Age, Customized [Count of Participants; unit: Participants]
  < 20 years | 2 | 2 | 16 | 10 | 30
  20-24 years | 16 | 14 | 34 | 42 | 106
  25-29 years | 20 | 16 | 30 | 26 | 92
  30-34 years | 4 | 6 | 12 | 16 | 38
  35+ years | 9 | 11 | 8 | 6 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 49 | 100 | 100 | 300
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 51 | 49 | 100 | 100 | 300
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Malawi | 51 | 49 | 100 | 100 | 300
Education [Count of Participants; unit: Participants]
  Primary school completed | 29 | 28 | 48 | 56 | 161
  Did not complete primary school | 22 | 21 | 52 | 44 | 139
Gestational age at enrollment, continuous [Median (Inter-Quartile Range); unit: weeks] | 26 [20 to 29] | 24 [19 to 28] | 28 [20 to 33] | 26 [17 to 34] | 26 [19.5 to 31]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Retained in Care With HIV Viral Suppression <40 Copies/mL (Groups 1a and 1b Only)
Description: The primary outcome measure is retention in care with HIV viral suppression, defined as <40 copies/mL.
Time Frame: 6 months following study enrollment
Population: Pregnant women living with HIV (Groups 1a and 1b only)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a: iNSC and Adherence Supporter Training | Group 1b: Standard of Care | Group 2a: iNSC and Adherence Supporter Training | Group 2b: Standard of Care
Number analyzed (Participants) | 51 | 49 | 0 | 0
Participants | 35 | 30 |  |

2. Primary Outcome: Number of Participants Retained in Care With Functional Adherence to PrEP (Groups 2a and 2b Only)
Description: The primary outcome is retention in care with functional adherence to PrEP as measured categorically according to plasma and intracellular tenofovir drug concentrations.
Time Frame: 6 months following study enrollment
Population: Pregnant women who are HIV-negative (Groups 2a and 2b only)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a: iNSC and Adherence Supporter Training | Group 1b: Standard of Care | Group 2a: iNSC and Adherence Supporter Training | Group 2b: Standard of Care
Number analyzed (Participants) | 0 | 0 | 100 | 100
Participants |  |  | 22 | 26

3. Secondary Outcome: Fidelity Score Indicating How Counselors Correctly Delivered Integrated Next Step Counseling by Session
Description: Extent to which Integrated Next Step Counseling (iNSC) was delivered as intended for each counseling session, obtained by audits of recorded counseling sessions. Counseling sessions were assessed according 50 evaluable actions. Each of these could be scored 0 (not done), 1 (partially done), and 2 (done well). These were aggregated into an overall score for fidelity, with an overall score range of 0-100. Higher scores represented greater counselor adherence to the iNSC framework.
Time Frame: 6 months following study enrollment
Population: Population comprises those in Groups 1a and 2a who attended their six month study visit and had a recorded counseling session for the visit
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Group 1a: iNSC and Adherence Supporter Training | Group 1b: Standard of Care | Group 2a: iNSC and Adherence Supporter Training | Group 2b: Standard of Care
Number analyzed (Participants) | 39 | 0 | 86 | 0
score on a scale | 89.3 [72.9 to 92.9] |  | 80.4 [70.7 to 86.4] |

4. Secondary Outcome: Reported Level of Satisfaction by Participants for the Study Intervention
Description: Satisfaction with overall intervention. Participants were asked: "How satisfied would you say you are with the program overall (both the iNSC and the Adherence Supporter)?" The five possible answers are shown below.
Time Frame: 6 months following study enrollment
Population: Satisfaction with the intervention measured only in those randomized to receive the intervention (Groups 1a and 2a)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a: iNSC and Adherence Supporter Training | Group 1b: Standard of Care | Group 2a: iNSC and Adherence Supporter Training | Group 2b: Standard of Care
Number analyzed (Participants) | 51 | 0 | 100 | 0
Participants
  Very satisfied | 42 |  | 89 |
  Somewhat satisfied | 1 |  | 2 |
  Neither satisfied nor unsatisfied | 0 |  | 0 |
  Somewhat unsatisfied | 0 |  | 0 |
  Very unsatisfied | 0 |  | 0 |
  Missing | 8 |  | 9 |

5. Secondary Outcome: Number of Participants Retained in Care With HIV Viral Suppression <1000 Copies/mL (Groups 1a and 1b Only)
Description: The secondary outcome measure is retention in care with HIV viral suppression, defined as <1000 copies/mL.
Time Frame: 6 months following study enrollment
Population: Pregnant women living with HIV (Groups 1a and 1b only)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a: iNSC and Adherence Supporter Training | Group 1b: Standard of Care | Group 2a: iNSC and Adherence Supporter Training | Group 2b: Standard of Care
Number analyzed (Participants) | 51 | 49 | 0 | 0
Participants | 37 | 35 |  |

6. Secondary Outcome: Number of Participants Retained in Care With ART Adherence >95% Over the Last 30 Days (Groups 1a and 1b Only)
Description: The secondary outcome measure is retention in care with self-reported ART adherence >95% over the last 30 days. Participants were asked how many pills they missed in the prior 30 days and this was used to calculate percent adherence, which was then dichotomized.
Time Frame: 6 months following study enrollment
Population: Pregnant women living with HIV (Groups 1a and 1b only)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a: iNSC and Adherence Supporter Training | Group 1b: Standard of Care | Group 2a: iNSC and Adherence Supporter Training | Group 2b: Standard of Care
Number analyzed (Participants) | 51 | 49 | 0 | 0
Participants | 37 | 32 |  |

7. Secondary Outcome: Number of Participants Retained in Care With >95% Adherence to PrEP Over Last 30 Days (Groups 2a and 2b Only)
Description: The secondary outcome is retention in care with >95% adherence to PrEP over the last 30 days by participant self-report. Participants were asked how many pills they missed in the prior 30 days and this was used to calculate percent adherence, which was then dichotomized.
Time Frame: 6 months following study enrollment
Population: Pregnant women who are HIV-negative (Groups 2a and 2b only)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a: iNSC and Adherence Supporter Training | Group 1b: Standard of Care | Group 2a: iNSC and Adherence Supporter Training | Group 2b: Standard of Care
Number analyzed (Participants) | 0 | 0 | 100 | 100
Participants |  |  | 45 | 43

8. Secondary Outcome: Number of Participants Reporting Social Harms
Description: Newly reported social harms during study follow-up period. At each study visit, participants were asked if they had encountered any social harms related to study participation. These were documented and, where appropriate, referrals to social services were made.
Time Frame: 3 months following study enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a: iNSC and Adherence Supporter Training | Group 1b: Standard of Care | Group 2a: iNSC and Adherence Supporter Training | Group 2b: Standard of Care
Number analyzed (Participants) | 51 | 49 | 100 | 100
Participants | 0 | 0 | 0 | 2

9. Secondary Outcome: Number of Participants Reporting Social Harms
Description: as for outcome 8
Time Frame: 6 months following study enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a: iNSC and Adherence Supporter Training | Group 1b: Standard of Care | Group 2a: iNSC and Adherence Supporter Training | Group 2b: Standard of Care
Number analyzed (Participants) | 51 | 49 | 100 | 100
Participants | 0 | 0 | 1 | 2

ADVERSE EVENTS:
Time Frame: From study enrollment through follow-up at 6 months (study visit window of 152 to 234 days).
Arm/Group | Group 1a: iNSC and Adherence Supporter Training | Group 1b: Standard of Care | Group 2a: iNSC and Adherence Supporter Training | Group 2b: Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/49 | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 4/51 | 2/49 | 11/100 | 6/100
Other Adverse Events (participants affected / at risk) | 1/51 | 7/49 | 5/100 | 6/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1a: iNSC and Adherence Supporter Training (N=51) | Group 1b: Standard of Care (N=49) | Group 2a: iNSC and Adherence Supporter Training (N=100) | Group 2b: Standard of Care (N=100)
Fetal demise (stillbirths and spontaneous abortions) (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 0 (0) | 8 (8) | 3 (3)
Neonatal death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Incident HIV infection (maternal) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — This applies only to Groups 2a and 2b.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1a: iNSC and Adherence Supporter Training (N=51) | Group 1b: Standard of Care (N=49) | Group 2a: iNSC and Adherence Supporter Training (N=100) | Group 2b: Standard of Care (N=100)
Preterm birth (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 7 (7) | 5 (5) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT04330989/Prot_SAP_000.pdf